CLINICAL TRIAL: NCT04441658
Title: Efficacy and Safety of Umbilical Cord Mesenchymal Stem Cells Transplantation in Patients With Type 2 Diabetes Mellitus
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai East Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DFSC-2020(CR)-02
Record Dates: First submitted 2020-06-19; First posted 2020-06-22 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Type 2 Diabetes; Mesenchymal Stem Cells
Keywords: Umbilical Cord Mesenchymal Stem Cells; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): The volunteers of the experimental group will be given peripheral intravenously a dose of 0.75*10^6/ kg human umbilical cord mesenchymal stem cells at 0,1,5,6 week.
  Interventions: Biological: Umbilical Cord Mesenchymal Stem Cells
- control group (Placebo Comparator): The control group will be given the same dose of saline containing human albumin.
  Interventions: Biological: saline

INTERVENTIONS:
Biological: Umbilical Cord Mesenchymal Stem Cells — human umbilical cord mesenchymal stem cells were peripheral intravenous infused to experimental group
  Arms: experimental group
Biological: saline — saline containing human albumin will be infused to the control group
  Arms: control group

SUMMARY:
This study is a 24-week single-center, randomized, double-blind, placebo-controlled trial. The trial includes a 3-week early screening and lifestyle education period, 6-week treatment period, and 18-week follow-up period. Chinese type 2 diabetic subjects receiving traditional hypoglycemic treatment were randomly assigned to umbilical cord mesenchymal stem cell or placebo infusion therapy to observe the efficacy and safety of umbilical cord mesenchymal stem cell infusion therapy.

DETAILED DESCRIPTION:
This study is a 24-week single-center, randomized, double-blind, placebo-controlled trial. The trial includes a 3-week early screening and lifestyle education period, 6-week treatment period, and 18-week follow-up period. Chinese type 2 diabetic subjects receiving traditional hypoglycemic treatment（including insulin） were randomly assigned to umbilical cord mesenchymal stem cell or placebo infusion therapy to observe the efficacy and safety of umbilical cord mesenchymal stem cell infusion therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes；
2. The course of diabetes is 5-15 years;
3. 20kg/m2≤body mass index (BMI)≤30 kg /m2；
4. 7.5% ≤HbA1c≤10%；
5. Insulin dose and other oral antidiabetic drugs doses should be stable over the 3 months prior to randomization.

Exclusion Criteria:

1. Heavy allergic constitution or an allergy to any component used in cell culture.
2. Being treated with drug (Glucocorticoids，Tricyclic Antidepressive Agents,etc.) affect the metabolism of glucose in the past 1 month;
3. other causes of diabetes;
4. All kinds of acute complications such as diabetic ketoacidosis and non-ketohyperosmotic syndrome were screened in the past 6 months;
5. Having evidence of ongoing or frequent/severe hypoglycemia in the past 6 months;
6. Severe cardiovascular and cerebral events：occurrence of heart failure NYHA Classification III or IV, myocardial infarction, cerebral infarction, cerebral hemorrhage within 6 months before the observation period;
7. Patients with abnormal liver and kidney function: AST and ALT exceeding 2.5 times of the normal upper limit, and serum creatinine exceeding 1.5 mg/dl for men, exceeding 1.4 mg/dl for women;
8. Positive results of HbsAg、Anti-HCV、HIV or syphilis;
9. Patients suffering from other serious systemic diseases (such as malignancy, central nervous system,cardiovascular system, blood system, digestive system,endocrine system,respiratory system, genitourinary system, immune system and);
10. Ongoing pregnancy or absence of effective contraception in women with childbearing potential;
11. Patients who had received other stem cell therapy before screening.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-04-10 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
The changes in HbA1C level | 24 weeks after treatment
  The changes in HbA1C level after transplantation

SECONDARY OUTCOMES:
Reduction of insulin requirement | 24 weeks after treatment
  Reduction of insulin requirement after transplantation
The changes in blood glucose level | 24 weeks after treatment
  The changes in blood glucose level after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: wang congrong, doctor, Principal Investigator — Shanghai East Hospital, China
Locations (1):
- Shanghai East Hospital, Shanghai Tongji University, Shanghai, Shanghai Municipality, China